CLINICAL TRIAL: NCT01555580
Title: A Pilot Study of Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) in Symptomatic Autoimmune Generalized Myasthenia Gravis
Brief Title: A Pilot Study of Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) in Generalized Myasthenia Gravis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Matthew N. Meriggioli, MD, Associate Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDA 2011 MG GM-CSF
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis; autoimmune; GM-CSF
MeSH Terms: conditions — Myasthenia Gravis | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GM-CSF (Experimental)
  Interventions: Drug: Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF)

INTERVENTIONS:
Drug: Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) — Participants will receive one dose of GM-CSF (5 µg/kg) by subcutaneous injection for ten (10) consecutive days. The first dose of GM-CSF will be administered by the subject or caregiver under the observation and direction of the study staff during the baseline visit. The subject or caregiver will administer subsequent injections at home.
  Other Names: LEUKINE® (sargramostim)

SUMMARY:
The purpose of this study is to determine whether the drug Leukine (GM-CFS) is safe and tolerated by patients with autoimmune myasthenia gravis (MG).

DETAILED DESCRIPTION:
Twelve patients aged 18-80 with symptomatic generalized autoimmune MG that are not being treated with medication that suppresses their immune system, other than prednisone, will enter the study at UIC over a two year period. The study will involve a screening visit and visits at baseline and at days 5, 15, 30, 45, 60, 90, and 120. The study drug, Leukine (GM-CFS), is given by injection. Subjects will give themselves one dose of GM-CSF every day for 10 days. Study visits will include muscle testing, immunologic studies and quality-of-life studies.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 80 years of age
* Established diagnosis of myasthenia based on: the presence of fatigable weakness of ocular, oropharyngeal, and/or limb muscles AND the presence of abnormal acetylcholine receptor binding antibodies ≥ 0.4 nmol/l.
* Patients of childbearing potential must agree to use a medically acceptable form of contraception defined by consistent use of oral contraceptive medications or history of tubal ligation or men who are in sexual relationship with such women during and for at least 8 weeks following completion of the study.
* Patient or designee must have the ability to self-inject investigational product
* If thymectomized, the procedure must have been performed at least one year prior to screening.
* Dose of current anticholinesterase drugs must be constant for 2 weeks prior to screening.
* If taking prednisone, dose must be stable for ≥4 weeks prior to screening.

Exclusion criteria:

* exclusively ocular MG (MGFA Class I)
* severe respiratory and/ or swallowing muscle weakness (MGFA Class Vb or V)
* presence of thymoma
* Must not have received plasm exchange or IVIG within 4 weeks of screening
* Must not have received immuno-modulating agents within the 4 weeks of screening, including Azathioprine (Imuran), Cyclosporine (Sandimmune, Neoral), Mycophenolate mofetil (CellCept), GM-CSF (Filgrastim; Neupogen; pegfilgrastim, sargramostim), or any other chronic immunosuppressive agent
* History of tuberculosis or evidence of latent tuberculosis (positive PPD skin test or a chest X-ray with evidence of tuberculosis)
* vital capacity of less than 1.2 liters or on supplemental oxygen therapy.
* severe comorbidities including lung disease, stroke, congestive heart failure of any severity, myocardial infarction, EKG abnormalities, uncontrolled hypertension - (sitting systolic BP <80 or > 160 mm Hg or diastolic BP > 100 mm Hg, unstable angina pectoris, hepatic or renal disease, insulin-dependent diabetes mellitus, history of cancer (other than in-situ cervical cancer or resected, cutaneous basal cell or squamous cell carcinoma), open cutaneous ulcers, known hepatitis B surface antigen (HbsAg) or hepatitis C virus (HCV) positive, or any other concurrent medical condition, which would make it unsafe for subjects to participate in the trial or interfere with the interpretation of the results.
* Laboratories values which, at the time of the screening visit or at any time during the study that in the opinion of the Investigator would preclude participation in the study including: serum creatinine > 2.5 mg/dL, serum potassium < 3.5 mmol/L or > 5.5 mmol/L, serum aspartate transaminase (AST), alanine transaminase (ALT), or alkaline phosphatase (ALP)> 3 times the upper limit of normal, platelet count < 100,000/mm3, WBC count < 3,000 cells/mm3, Hemoglobin, hematocrit, or red blood cell count outside 30% of the upper or lower limits of normal
* Receipt of a live vaccine within 3 months of screening
* participation in another investigational drug study within 90 days of screening.
* known hypersensitivity to GM-CSF or any of its components
* Known HIV-positive status or known history of any other immuno-suppressing disease.
* Any mycobacterial disease.
* Active severe infections within 4 weeks before screening visit, or between the screening and baseline visits.
* Untreated Lyme disease.
* History of TB or TB exposure, chronic hepatitis B or hepatitis C, SLE, history of multiple sclerosis, transverse myelitis, optic neuritis or epilepsy.
* History of recent alcohol or substance abuse (< 1 year)
* Pregnant or lactating females
* History of non-compliance with other therapies
* abnormal mental status sufficient to exclude informed consent
* History of any opportunistic infection - to include but not limited to Pneumocystis carinii, aspergillosis, histoplasmosis, or atypical mycobacterium
* History of Sickle cell disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety of GM-CSF in patients with myasthenia gravis | 150 days
  The number of subjects experiencing a Class II-V adverse event within 120 days of the start of treatment that is probably or definitely related to the study medication
The change from baseline in the quantitative and functional (suppressive capacity) characterization of circulating regulatory T cells at 30 days post-treatment | 30 days
The change from baseline in the quantitative and functional (suppressive capacity) characterization of circulating regulatory T cells at 60 days post-treatment | 60 days
The change from baseline in the quantitative and functional (suppressive capacity) characterization of circulating regulatory T cells at 120 days post-treatment | 120 days

SECONDARY OUTCOMES:
Change from baseline in the Quantitative Myasthenia Gravis (QMG) score at 60 days | 60 days
Change from baseline in the Quantitative Myasthenia Gravis (QMG) score at day 120 | 120 days
Change from baseline in the Myasthenia Gravis Composite score at day 60 | 60 days
Change from baseline in the Myasthenia Gravis Composite score at day 120 | 120 days
Change from baseline in Manual Muscle Testing (MMT) score at day 60 | 60 days
Change from baseline in Manual Muscle Testing (MMT) score at day 120 | 120 days
Change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) score at day 60 | 60 days
Change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) score at day 120 | 120 days
Change from baseline in Quality of Life Assessment (SF-36) at day 60 | 60 days
Change from baseline in Quality of Life Assessment (SF-36) at day 120 | 120 days
Change from baseline in acetylcholine receptor antibody titre level at day 60 | 60 days
Change from baseline in acetylcholine receptor antibody titre level at day 120 | 120 days
Change from baseline in prednisone dose at day 60 | 60 days
Change from baseline in prednisone dose at day 120 Days | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew N Meriggioli, MD, Principal Investigator — University of Illinois at Chicago, 912 S. Wood St., Rm 855-N, M/C 796, Chicago IL 60612
Locations (1):
- University of Illinois at Chicago, Department of Neurology, Chicago, Illinois, United States